CLINICAL TRIAL: NCT06257940
Title: Impact of Changing Sterile Glove at the Time of Wound Closure to Reduce Surgical Site Infection in Women Undergoing Elective Cesarean Section; a Prospective Randomized Controlled Clinical Trial
Brief Title: Impact of Changing Sterile Glove at the Time of Wound Closure to Reduce Surgical Site Infection
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naglaa Hamada Mohamed, doctor, Assiut University
Other Study IDs: 04-2023-200359
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intra-operative glove changing group: in which, the surgeon will replace his/her outer surgical gloves with a new pair of sterile gloves just prior to abdominal closure
- usual care group: in which, surgeon won't change his/her gloves before abdominal closure

SUMMARY:
Assessment of the impact of changing sterile gloves at the time of wound closure on reduction of SSI in women undergoing elective CS.

DETAILED DESCRIPTION:
1. CS is the most common major operation preformed worldwide. In daily obstetric practice. It account for up to 60% of all births in some countries .
2. Previous study reported that Egypt has the third highest CS rate (54%) in the world and lacks a standard classification system to analyze CS rates, following Do-minican Republic (56.4 percent) and Brazil (55.6 percent). Within the Arab region, rates of CS are far higher in Egypt than any other Arab country .
3. In another study, the CS rate in Egypt was estimated at 55.1%, and the highest rate was 67.8% in Behira and the lowest was 49.0% in Assiut. In most governorates, the CS rate was higher in rural than in urban areas, but the difference was not significant. High CS rates were significantly related to higher social class and lower number of children (≤ 3).
4. The percentage of "unjustified" caesarean deliveries has exceeded 62 percent of total deliveries in Egypt, many of which could have been done naturally. In August 2022, the Central Agency for Public Mobilization and Statistics (CAPMAS) reported a noticeable increase in C-sections in recent years. CAPMAS found that C-sections increased to 72 percent of all deliveries in 2021, up from 52 percent in 2014. The agency also found that C-sections in rural areas increased to 84 percent of all deliveries in 2021, up from 70.6 percent in 2014.
5. One of the most serious complications after CS is wound complication it varies from 3 to 30% .
6. It may be infectious as SSI or non-infectious as hematoma, seroma, and wound separation. These complications cause increase hospital stay or readmission also, maternal morbidaty and cost are increased .
7. SSIs are a common cause of health care-associated infection. The United States Centers for Disease Control and Prevention (CDC) has developed criteria that define SSI as infection related to an operative procedure that occurs at or near the surgical incision within 30 days of the procedure or within 90 days if prosthetic material is implanted at surgery. SSIs are often localized to the incision site (superficial/deep incisional SSI) but can also extend into deep tissues .
8. There were numerous recommendations for SSI prevention efforts in recent World Health Organization (WHO) guidelines, however most of these interventions were not well-supported by high-quality evidence .
9. WHO recommendations for change of gloves at the time of fascial closure were identified as the priority recommendations. Three studies have been published to date, all suggesting to a benefit, however the particular evidence for SSI reduction with glove change prior to fascial closure is limited, consisting primarily of small RCTs with a high risk of bias .
10. The CDC, WHO, and NICE guidelines do not recommend changing gloves as part of routine care due to the poor evidence data base. The executive summary of the 2017 WHO Guidelines on SSI Reduction Practice indicates that well-designed RCTs would be requested because there is no direct proof of the usefulness of sterile surgical gloves changing prior to wound closure .
11. The CDC healthcare-associated infection (HAI) prevalence survey found that there were an estimated 110,800 SSIs associated with inpatient surgeries in 2015. SSI is the most costly HAI type with an estimated annual cost of $3.3 billion, and extends hospital length of stay by 9.7 days, with cost of hospitalization increased by more than $20,000 per admission

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-35 years.
* Non obese with body mass index (BMI) < 30 kg/m2.
* Term pregnancy ≥ 37 weeks +0 days.
* Singleton.
* Viable fetus.

Exclusion Criteria:

* Obese women with body mass index (BMI) ≥ 30 kg/m2.
* Anemic women with hemoglobin level < 10.5 g/dl.
* Immuno-compromised women with medical disorders with pregnancy as diabetes mellitus, hypertension, cardiac, hepatic or renal disorders.
* Women with anticipated pelvic adhesions as cases with history of endometriosis, pelvic inflammatory diseases or more than previous 3 CSs.
* Multifetal pregnancy.
* Emergency CS.
* Women with antepartum hemorrhage (placenta previa or placenta accrete spectrum disorder).
* Obstetric cases with increased risk of infection as premature rapture of membranes (PROMs).
* Women refusing to participate in the study.

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: study will be conducted in Assuit Women Health Hospital We will recruit a pregnant women attending for cesarean sections according to the previous inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Changing Sterile Glove at the Time of Wound Closure to Reduce Surgical Site Infection | within 4 weeks after cesarean sections
  Composite end point of any wound complication i.e. SSI occurring within one and three weeks following delivery. These wound complications include wound seroma, wound hematoma, wound infection, skin separation of at least 1 cm or other incisional abnormality requiring a bedside procedure to treat.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abu El-Fadl El-Sayed, assistant professor, Study Director — obstetrics & gynacology depatmen assiut university
Locations (1):
- assiut University, Asyut, Egypt

REFERENCES:
- [Background] Wahdan M, Hakim S, El Gaafary M, Sos D, Wassif G, Hussein W, Mokhtar A, Hussein A, El Awady M, Rady M, Anwar W. Rising trends in Caesarean section in 6 Egyptian governorates. East Mediterr Health J. 2022 May 29;28(5):336-344. doi: 10.26719/emhj.22.012. PMID 35670438
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Kawakita T, Landy HJ. Surgical site infections after cesarean delivery: epidemiology, prevention and treatment. Matern Health Neonatol Perinatol. 2017 Jul 5;3:12. doi: 10.1186/s40748-017-0051-3. eCollection 2017. PMID 28690864
- [Background] Ban KA, Minei JP, Laronga C, Harbrecht BG, Jensen EH, Fry DE, Itani KM, Dellinger EP, Ko CY, Duane TM. American College of Surgeons and Surgical Infection Society: Surgical Site Infection Guidelines, 2016 Update. J Am Coll Surg. 2017 Jan;224(1):59-74. doi: 10.1016/j.jamcollsurg.2016.10.029. Epub 2016 Nov 30. No abstract available. PMID 27915053